CLINICAL TRIAL: NCT00700336
Title: Phase I/II Study of a Triplet Combination of CBP501, Pemetrexed and Cisplatin in Patients With Advanced Solid Tumors and in Chemotherapy-naïve Patients With Malignant Pleural Mesothelioma
Brief Title: Study of CBP501 + Pemetrexed + Cisplatin on MPM (Phase I/II)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CanBas Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBP08-01
Record Dates: First submitted 2008-06-16; First posted 2008-06-18 (Estimated); Results first posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-06

CONDITIONS: Malignant Pleural Mesothelioma; Solid Tumors
Keywords: malignant pleural mesothelioma; solid tumors
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Pemetrexed; Cisplatin; Cdc25C phosphatase (211-221)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pemetrexed, Cisplatin, and CBP501: Phase 2 (Experimental): pemetrexed, cisplatin and CBP501
  Interventions: Drug: pemetrexed, cisplatin and CBP501
- Pemetrexed and Cisplatin: Phase 2 (Active Comparator): pemetrexed and cisplatin
  Interventions: Drug: pemetrexed and cisplatin
- Pemetrexed, Cisplatin, and CBP501:Phase 1 (Experimental): MTD, which was equal to recommended dose for the Phase II part, was determined by 6 patients (3+3)
  Interventions: Drug: pemetrexed, cisplatin and CBP501, dose finding

INTERVENTIONS:
Drug: pemetrexed, cisplatin and CBP501 — CBP501 25 mg/m2, Pemetrexed 500 mg/m2, cisplatin 75 mg/m2 CBP501 for injection is provided in single dose vials (20 mg) containing a sterile lyophilized powder comprising CBP501 peptide acetate salt (peptide base units). For administration, vial contents are reconstituted in 5% Dextrose Injection, USP, and added to a 100 mL IV bag of 5% Dextrose Injection, USP.
  Pemetrexed: A commercial formulation of pemetrexed will be used, with reconstitution in 20mL 0.9% sodium chloride solution for injection, then dilution to 100mL.
  Cisplatin: A commercial formulation will be used and will be diluted in 250 mL of normal saline for administration.
  Other Names: Arm A
  Arms: Pemetrexed, Cisplatin, and CBP501: Phase 2
Drug: pemetrexed and cisplatin — Pemetrexed 500 mg/m2, cisplatin 75 mg/m2 Pemetrexed: A commercial formulation of pemetrexed will be used, with reconstitution in 20mL 0.9% sodium chloride solution for injection, then dilution to 100mL.
  Cisplatin: A commercial formulation will be used and will be diluted in 250 mL of normal saline for administration.
  Other Names: Arm B
  Arms: Pemetrexed and Cisplatin: Phase 2
Drug: pemetrexed, cisplatin and CBP501, dose finding — Dose level 1: CBP501 16 mg/m2, Pemetrexed 500 mg/m2, cisplatin 75 mg/m2 Dose level 2: CBP501 25 mg/m2, Pemetrexed 500 mg/m2, cisplatin 75 mg/m2 CBP501 for injection is provided in single dose vials (20 mg) containing a sterile lyophilized powder comprising CBP501 peptide acetate salt (peptide base units). For administration, vial contents are reconstituted in 5% Dextrose Injection, USP, and added to a 100 mL IV bag of 5% Dextrose Injection, USP.
  Pemetrexed: A commercial formulation of pemetrexed will be used, with reconstitution in 20mL 0.9% sodium chloride solution for injection, then dilution to 100mL.
  Cisplatin: A commercial formulation will be used and will be diluted in 250 mL of normal saline for administration.
  Other Names: Phase I part; Dose finding
  Arms: Pemetrexed, Cisplatin, and CBP501:Phase 1

SUMMARY:
The phase I part of the study is a dose-finding study of escalating doses of CBP501 combined with full-dose cisplatin and pemetrexed in patients with histologically confirmed solid malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective or would otherwise be eligible for cisplatin and pemetrexed as first-line therapy. The maximum tolerated dose (MTD) will be determined based on DLTs occurring during the first treatment cycle. Pharmacokinetics of the triplet combination will be assessed during the phase I part of the trial.

The phase II part will evaluate full-dose cisplatin and pemetrexed combined with CBP501 (at the MTD determined in the phase I part) in previously untreated, unresectable malignant pleural mesothelioma patients. Patients will be randomized in a 2 : 1 ratio to pemetrexed, cisplatin and CBP501 (Arm A) or to pemetrexed and cisplatin (Arm B); randomization will be stratified according to histology and performance status.

DETAILED DESCRIPTION:
This is an open-label, multicenter, international, phase I-II study. The phase I part, a dose-finding study of escalating doses of CBP501 combined with fixed full-dose cisplatin and pemetrexed, has been completed and results are presented in this report. MTD was determined on DLT occurring during the first cycle. This phase I part was evaluated in a patient population with advanced solid tumors The phase II part will evaluate full-dose cisplatin and pemetrexed combined with CBP501 at the MTD determined in the phase I part. Patients will be randomized in a 2:1 ratio to pemetrexed, cisplatin and CBP501 (Arm A) or pemetrexed and cisplatin (Arm B). This phase II part will be evaluated in chemotherapy-naïve patients with malignant pleural mesothelioma

Randomization will be stratified by:

* Histology: epithelial vs other (sarcomatoid or biphasic)
* Performance status: 0-1 vs 2

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent obtained prior to initiation of any study-specific procedures
2. Phase I: Histologically confirmed solid malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective or would otherwise be eligible for cisplatin and pemetrexed as first-line therapy

   Phase II: Histologically or cytologically confirmed diagnosis of malignant pleural mesothelioma (MPM), not amenable for radical resection, who has not received previous chemotherapy or other systemic treatment
3. Measurable disease according to the modified Response Evaluation Criteria in Solid Tumors (RECIST, see below)
4. Male or female patients aged at least 18 years
5. ECOG Performance Status (PS): 0-2
6. Previous anticancer treatment must be discontinued at least 3 weeks prior to first dose of study treatment (6 weeks for mitomycin C; 6 weeks for anti-androgen therapy if discontinued prior to treatment initiation, with the exception of 8 weeks for bicalutamide)
7. Life expectancy greater than 3 months
8. Adequate organ function
9. Female patients of child-bearing potential must have a negative pregnancy test and be using at least one form of contraception as approved by the Investigator for 4 weeks prior to the study and 4 months after the last dose of study drug. For the purposes of this study, child-bearing potential is defined as: "All female patients unless they are post-menopausal for at least one year or are surgically sterile"
10. Male patients must use a form of barrier contraception approved by the investigator during the study and for 4 months after the last dose of study drug
11. Ability to cooperate with the treatment and follow-up

Exclusion Criteria:

1. Radiation therapy to more than 30% of the bone marrow prior to entry into the study
2. Phase II only: Mesothelioma originating outside the pleura (e.g.: peritoneum)
3. Absence of measurable lesions
4. The patient has an ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, symptomatic or poorly controlled cardiac arrhythmia, uncontrolled thrombotic or hemorrhagic disorder, or any other serious uncontrolled medical disorders in the opinion of the investigator.
5. Any previous history of another malignancy within 5 years of study entry (other than cured basal cell carcinoma of the skin or cured in-situ carcinoma of the cervix)
6. Presence of any significant central nervous system or psychiatric disorder(s) that would hamper the patient's compliance
7. Evidence of peripheral neuropathy > grade 1 according to NCI-CTCAE Version 3
8. Treatment with any other investigational agent, or participation in another clinical trial within 28 days prior to study entry
9. Pregnant or breast-feeding patients or any patient with childbearing potential not using adequate contraception
10. Known HIV, HBV, HCV infection
11. Presence of CNS metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2008-05; Primary Completion 2012-07 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Krug, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (12):
- United States (12):
  - Mayo Clinic, Scottsdale, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - City of Hope, Duarte, California
  - University of Chicago, Chicago, Illinois
  - Karmanos Cancer Institute/Wayne State University, Detroit, Michigan
  - Nevada Cancer Institute, Las Vegas, Nevada
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial-Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Penn State Milton S. Hershey Medical Ctr., Hershey, Pennsylvania
  - Cancer Therapy & Research Center, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suganuma M, Kawabe T, Hori H, Funabiki T, Okamoto T. Sensitization of cancer cells to DNA damage-induced cell death by specific cell cycle G2 checkpoint abrogation. Cancer Res. 1999 Dec 1;59(23):5887-91. PMID 10606229
- [Background] Sha SK, Sato T, Kobayashi H, Ishigaki M, Yamamoto S, Sato H, Takada A, Nakajyo S, Mochizuki Y, Friedman JM, Cheng FC, Okura T, Kimura R, Kufe DW, Vonhoff DD, Kawabe T. Cell cycle phenotype-based optimization of G2-abrogating peptides yields CBP501 with a unique mechanism of action at the G2 checkpoint. Mol Cancer Ther. 2007 Jan;6(1):147-53. doi: 10.1158/1535-7163.MCT-06-0371. PMID 17237275
- [Background] Mine N, Yamamoto S, Saito N, Yamazaki S, Suda C, Ishigaki M, Kufe DW, Von Hoff DD, Kawabe T. CBP501-calmodulin binding contributes to sensitizing tumor cells to cisplatin and bleomycin. Mol Cancer Ther. 2011 Oct;10(10):1929-38. doi: 10.1158/1535-7163.MCT-10-1139. Epub 2011 Aug 10. PMID 21831962
- [Background] Shapiro GI, Tibes R, Gordon MS, Wong BY, Eder JP, Borad MJ, Mendelson DS, Vogelzang NJ, Bastos BR, Weiss GJ, Fernandez C, Sutherland W, Sato H, Pierceall WE, Weaver D, Slough S, Wasserman E, Kufe DW, Von Hoff D, Kawabe T, Sharma S. Phase I studies of CBP501, a G2 checkpoint abrogator, as monotherapy and in combination with cisplatin in patients with advanced solid tumors. Clin Cancer Res. 2011 May 15;17(10):3431-42. doi: 10.1158/1078-0432.CCR-10-2345. Epub 2011 Jan 10. PMID 21220472
- [Background] Matsumoto Y, Shindo Y, Takakusagi Y, Takakusagi K, Tsukuda S, Kusayanagi T, Sato H, Kawabe T, Sugawara F, Sakaguchi K. Screening of a library of T7 phage-displayed peptides identifies alphaC helix in 14-3-3 protein as a CBP501-binding site. Bioorg Med Chem. 2011 Dec 1;19(23):7049-56. doi: 10.1016/j.bmc.2011.10.004. Epub 2011 Oct 7. PMID 22032894

RESULTS

PARTICIPANT FLOW:
Groups:
- Pemetrexed, Cisplatin and CBP501: Phase 2: pemetrexed, cisplatin and CBP501: CBP501 for injection is provided in single dose vials (20 mg) containing a sterile lyophilized powder comprising CBP501 peptide acetate salt (peptide base units). For administration, vial contents are reconstituted in 5% Dextrose Injection, USP, and added to a 100 mL IV bag of 5% Dextrose Injection, USP.
  Pemetrexed: A commercial formulation of pemetrexed will be used, with reconstitution in 20mL 0.9% sodium chloride solution for injection, then dilution to 100mL.
  Cisplatin: A commercial formulation will be used and will be diluted in 250 mL of normal saline for administration.
- Pemetrexed and Cisplatin: Phase 2: pemetrexed and cisplatin: Pemetrexed: A commercial formulation of pemetrexed will be used, with reconstitution in 20mL 0.9% sodium chloride solution for injection, then dilution to 100mL.
  Cisplatin: A commercial formulation will be used and will be diluted in 250 mL of normal saline for administration.
- Pemetrexed, Cisplatin and CBP501: Phase 1: DL1: CBP501 16mg/m2, pemetrexed 500mg/m2, cisplatin 75mg/m2 DL2: CBP501 25mg/m2, pemetrexed 500mg/m2, cisplatin 75mg/m2
Period: Overall Study
Arm/Group | Pemetrexed, Cisplatin and CBP501: Phase 2 | Pemetrexed and Cisplatin: Phase 2 | Pemetrexed, Cisplatin and CBP501: Phase 1
Started | 40 | 23 | 6
Completed | 40 | 23 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pemetrexed, Cisplatin, and CBP501: Phase 2: pemetrexed, cisplatin and CBP501
  pemetrexed, cisplatin and CBP501: CBP501 for injection is provided in single dose vials (20 mg) containing a sterile lyophilized powder comprising CBP501 peptide acetate salt (peptide base units). For administration, vial contents are reconstituted in 5% Dextrose Injection, USP, and added to a 100 mL IV bag of 5% Dextrose Injection, USP.
  Pemetrexed: A commercial formulation of pemetrexed will be used, with reconstitution in 20mL 0.9% sodium chloride solution for injection, then dilution to 100mL.
  Cisplatin: A commercial formulation will be used and will be diluted in 250 mL of normal saline for administration.
- Pemetrexed and Cisplatin: Phase 2: pemetrexed and cisplatin
  pemetrexed and cisplatin: Pemetrexed: A commercial formulation of pemetrexed will be used, with reconstitution in 20mL 0.9% sodium chloride solution for injection, then dilution to 100mL.
  Cisplatin: A commercial formulation will be used and will be diluted in 250 mL of normal saline for administration.
- Pemetrexed, Cisplatin, and CBP501: Phase 1: DL1: CBP501 16mg/m2, Alimta 500mg/m2, cisplatin 75mg/m2 DL2: CBP501 25mg/m2, Alimta 500mg/m2, cisplatin 75mg/m2
- Total: Total of all reporting groups
Arm/Group | Pemetrexed, Cisplatin, and CBP501: Phase 2 | Pemetrexed and Cisplatin: Phase 2 | Pemetrexed, Cisplatin, and CBP501: Phase 1 | Total
Number analyzed (Participants) | 40 | 23 | 6 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (10.03) | 66.3 (12.10) | 62.8 (13.61) | 64.2 (10.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 1 | 12
  Male | 32 | 20 | 5 | 57

OUTCOME MEASURES:

1. Primary Outcome: 4M PFS Rate of Patients With Previously Untreated, Unresectable Malignant Pleural Mesothelioma (MPM) Treated With CBP501, Pemetrexed and Cisplatin
Description: Planned: Forty-two patients were to be treated in Arm A. If ≥ 23 patients (>54%) were free of progression and death at 4 months, then the study regimen would be considered for further evaluation in this indication.
Time Frame: End of study
Measure: Number; unit: participants
Groups:
- Pemetrexed, Cisplatin, and CBP501: Pemetrexed, Cisplatin, and CBP501 administered once every 3 weeks
- Pemetrexed and Cisplatin: Pemetrexed and Cisplatin every three weeks
Arm/Group | Pemetrexed, Cisplatin, and CBP501 | Pemetrexed and Cisplatin
Number analyzed (Participants) | 40 | 23
participants
  4M PFS by Independent Image Review | 25 | 9
  4M PFS by Site assess | 27 | 13

ADVERSE EVENTS:
Arm/Group | Pemetrexed, Cisplatin, and CBP501: Phase 2 | Pemetrexed and Cisplatin: Phase 2 | Pemetrexed, Cisplatin, and CBP501: Phase 1
All-Cause Mortality (participants affected / at risk) | 1/40 | 1/23 | 4/6
Serious Adverse Events (participants affected / at risk) | 21/40 | 13/23 | 5/6
Other Adverse Events (participants affected / at risk) | 28/40 | 15/23 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed, Cisplatin, and CBP501: Phase 2 (N=40) | Pemetrexed and Cisplatin: Phase 2 (N=23) | Pemetrexed, Cisplatin, and CBP501: Phase 1 (N=6)
Lymphopenia (Blood and lymphatic system disorders) | 2 | 1 | 0
abdominal pain (Gastrointestinal disorders) | 0 | 3 | 1
Nausea (Gastrointestinal disorders) | 3 | 2 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1 | 0
Fatigue (General disorders) | 7 | 3 | 0
Haemoglobin decreased (Investigations) | 3 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 4 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 2 | 0
Malignant neoplasm progressed (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
renal failure (Renal and urinary disorders) | 2 | 0 | 0
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
deep vein thrombosis (Vascular disorders) | 2 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Syncope (Vascular disorders) | 0 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed, Cisplatin, and CBP501: Phase 2 (N=40) | Pemetrexed and Cisplatin: Phase 2 (N=23) | Pemetrexed, Cisplatin, and CBP501: Phase 1 (N=6)
anemia (Blood and lymphatic system disorders) | 7 | 8 | 3
leukopenia (Blood and lymphatic system disorders) | 2 | 1 | 0
lymphopenia (Blood and lymphatic system disorders) | 5 | 1 | 0
neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 1
tinnitus (Ear and labyrinth disorders) | 5 | 2 | 0
lacrimation increased (Eye disorders) | 2 | 2 | 1
vision blurred (Eye disorders) | 2 | 0 | 1
abdominal discomfort (Gastrointestinal disorders) | 2 | 1 | 0
abdominal distension (Gastrointestinal disorders) | 1 | 3 | 2
abdominal pain (Gastrointestinal disorders) | 4 | 1 | 1
constipation (Gastrointestinal disorders) | 21 | 15 | 4
diarrhea (Gastrointestinal disorders) | 8 | 4 | 2
dry mouth (Gastrointestinal disorders) | 2 | 2 | 0
dyspepsia (Gastrointestinal disorders) | 5 | 2 | 1
nausea (Gastrointestinal disorders) | 24 | 13 | 5
stomatitis (Gastrointestinal disorders) | 2 | 1 | 3
vomiting (Gastrointestinal disorders) | 8 | 9 | 1
asthenia (General disorders) | 2 | 0 | 0
chest discomfort (General disorders) | 2 | 1 | 0
chest pain (General disorders) | 7 | 4 | 0
chills (General disorders) | 2 | 0 | 2
fatigue (General disorders) | 24 | 15 | 5
infusion related reactions (General disorders) | 28 | 0 | 2
infusion site rash (General disorders) | 2 | 0 | 0
mucosal inflammation (General disorders) | 2 | 1 | 0
oedema peripheral (General disorders) | 5 | 6 | 0
pain (General disorders) | 1 | 2 | 0
pyrexia (General disorders) | 6 | 3 | 1
hypersensitivity (Immune system disorders) | 0 | 2 | 0
oral candidiasis (Infections and infestations) | 2 | 0 | 0
blood albumin decreased (Investigations) | 2 | 0 | 0
blood creatinine increased (Investigations) | 7 | 3 | 1
blood glucose increased (Investigations) | 2 | 0 | 0
blood sodium decreased (Investigations) | 2 | 0 | 0
ECG QT prolonged (Investigations) | 2 | 1 | 1
hemoglobin decreased (Investigations) | 7 | 0 | 0
neutrophil count decreased (Investigations) | 2 | 0 | 0
platelet count decreased (Investigations) | 3 | 1 | 0
prothrombin time prolonged (Investigations) | 2 | 0 | 0
weight decreased (Investigations) | 5 | 1 | 0
WBC decreased (Investigations) | 4 | 0 | 0
decreased apetite (Metabolism and nutrition disorders) | 18 | 12 | 0
dehydration (Metabolism and nutrition disorders) | 6 | 2 | 0
hyperglycemia (Metabolism and nutrition disorders) | 4 | 2 | 0
hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 1 | 0
hypokalemia (Metabolism and nutrition disorders) | 2 | 1 | 0
hypomagnesemia (Metabolism and nutrition disorders) | 4 | 4 | 2
hyponatremia (Metabolism and nutrition disorders) | 3 | 2 | 1
arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 8 | 2 | 0
myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
dizziness (Nervous system disorders) | 2 | 2 | 2
dysgeusia (Nervous system disorders) | 7 | 3 | 0
Headache (Nervous system disorders) | 5 | 0 | 2
neurophaty peripheral (Nervous system disorders) | 7 | 3 | 3
peropheral sensory neuropathy (Nervous system disorders) | 1 | 3 | 0
anxiety (Psychiatric disorders) | 4 | 3 | 0
insomnia (Psychiatric disorders) | 2 | 3 | 3
renal failure (Renal and urinary disorders) | 1 | 2 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 7 | 11 | 5
dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 | 8 | 3
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
hiccups (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 2
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
alopecia (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
night sweats (Skin and subcutaneous tissue disorders) | 2 | 1 | 2
pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 2
rash (Skin and subcutaneous tissue disorders) | 9 | 1 | 2
hypertension (Vascular disorders) | 5 | 0 | 2
phlebitis (Vascular disorders) | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No